CLINICAL TRIAL: NCT03046576
Title: The Association Between Plasma DPP4 Activity And Prognosis of Patients With ST-Elevation Myocardial Infarction Undergoing Percutaneous Coronary Intervention
Brief Title: Prognostic Value of Plasma DPP4 Activity in ST-elevation Myocardial Infarction Patients
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Li Jing Wei, MD, Dr., Chinese PLA General Hospital
Other Study IDs: DPP4a-MACCE
Record Dates: First submitted 2017-02-05; First posted 2017-02-08 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Coronary Angiography; Dipeptidyl Peptidase 4

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: plasma DPP4 activity — DPP4a was determined by enzymatic assays.

SUMMARY:
Increased plasma DPP4 activity (DPP4a) could predict both subclinical and new-onset atherosclerosis, and our previous study has found that the DPP4a was significantly lower in MI patients compared with patients having chest pain or unstable angina alone, and DPP4a is associated with no-reflow and major bleeding events in STEMI patients during hospital stay. As no-reflow phenomenon and major bleeding events independently associates with a worse in-hospital and long-term prognosis. One may speculate that the DPP4a is associated with long-term follow-up adverse cardiovascular events in these patients.The hypothesis was tested in this study.

ELIGIBILITY:
Inclusion Criteria:

* consecutive patients of acute STEMI come to our department,absent of cardiogenic shock, and survival for at least 24 h after PCI treatment.

Exclusion Criteria:

* patients with cancer, and patients who were taking a DPP4 inhibitoror a glucagon-like peptide-1 (GLP-1) analogue

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with STEMI who were admitted to the Chinese PLA General Hospital for PCI
Sampling Method: Probability Sample
Enrollment: 625 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2015-09-30 (Actual); Study Completion 2015-09-30 (Actual)

PRIMARY OUTCOMES:
major adverse cardiac or cerebrovascular events | The median follow-up was 30 months
  including cardiovascular death, non-fatal myocardial infarction, heart failure and stroke

SECONDARY OUTCOMES:
non-cardiovascular death | The median follow-up was 30 months
repeated revascularization | The median follow-up was 30 months
  defined as repeated PCI or bypass grafting of not only infarct related artery but also non-infarct related artery, driven by ischemic symptoms (stable/unstable angina or re-infarction) or detection of ischemia by non-invasive tests
stroke | The median follow-up was 30 months
  defined using the World Health Organization criteria

REFERENCES:
- [Background] Zheng TP, Liu YH, Yang LX, Qin SH, Liu HB. Increased plasma dipeptidyl peptidase-4 activities are associated with high prevalence of subclinical atherosclerosis in Chinese patients with newly diagnosed type 2 diabetes: a cross-sectional study. Atherosclerosis. 2015 Oct;242(2):580-8. doi: 10.1016/j.atherosclerosis.2015.07.042. Epub 2015 Jul 26. PMID 26318108
- [Background] Zheng TP, Yang F, Gao Y, Baskota A, Chen T, Tian HM, Ran XW. Increased plasma DPP4 activities predict new-onset atherosclerosis in association with its proinflammatory effects in Chinese over a four year period: A prospective study. Atherosclerosis. 2014 Aug;235(2):619-24. doi: 10.1016/j.atherosclerosis.2014.05.956. Epub 2014 Jun 8. PMID 24968315
- [Background] Li JW, Chen YD, Chen WR, Jing J, Liu J, Yang YQ. Plasma DPP4 activity is associated with no-reflow and major bleeding events in Chinese PCI-treated STEMI patients. Sci Rep. 2016 Dec 21;6:39412. doi: 10.1038/srep39412. PMID 28000723
- [Background] Niccoli G, Kharbanda RK, Crea F, Banning AP. No-reflow: again prevention is better than treatment. Eur Heart J. 2010 Oct;31(20):2449-55. doi: 10.1093/eurheartj/ehq299. Epub 2010 Sep 13. No abstract available. PMID 20837571
- [Background] Pellaton C, Cayla G, Silvain J, Zeymer U, Cohen M, Goldstein P, Huber K, Pollack C Jr, Kerneis M, Collet JP, Vicaut E, Montalescot G; ATOLL Investigators. Incidence and consequence of major bleeding in primary percutaneous intervention for ST-elevation myocardial infarction in the era of radial access: an analysis of the international randomized Acute myocardial infarction Treated with primary angioplasty and intravenous enoxaparin Or unfractionated heparin to Lower ischemic and bleeding events at short- and Long-term follow-up trial. Am Heart J. 2015 Oct;170(4):778-86. doi: 10.1016/j.ahj.2015.05.021. Epub 2015 Jul 3. PMID 26386802
- [Derived] Li JW, Chen YD, Chen WR, You Q, Li B, Zhou H, Zhang Y, Han TW. Prognostic value of plasma DPP4 activity in ST-elevation myocardial infarction. Cardiovasc Diabetol. 2017 Jun 6;16(1):72. doi: 10.1186/s12933-017-0553-3. PMID 28587613